CLINICAL TRIAL: NCT01963455
Title: The Effect Evaluation of Autologous Muscle Derived Stem Cells Injection Into the Paraurethral Tissues for Treatment of Urinary Incontinency
Brief Title: Autologous Muscle Derived Stem Cells Transplantation in Urine Incontinency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: royan-Kidney-001
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2013-01

CONDITIONS: Stress Incontinency
Keywords: transplantation autologous stress urinary incontinence; muscle derived cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDCs transplant (Experimental): The women who have stress urinary incontinency.
  Interventions: Biological: paraurethral injection of MDCs

INTERVENTIONS:
Biological: paraurethral injection of MDCs — MDCs transplantation by paraurethral injection .
  Other Names: MDCs transplantion by paraurethral injection.

SUMMARY:
This study was designed to provide confirmation of safety of muscle derived cell (MDCs) for the treatment of stress urine incontinency (SUI) in women.

DETAILED DESCRIPTION:
The investigators will be assessed the 12-month safety and potential efficacy of autologous muscle derived cells as therapy for stress urinary incontinence. A total of 10 women in whom stress urinary incontinence had not improved underwent intra-sphincter injection of low doses 30×106 of autologous muscle derived cells, which will be derived from biopsies of their deltoid muscle. Assessments will be made at 1, 3, 6 and 12 months after cell injection. Changes in stress urinary incontinence severity were evaluated by pad test, diary of incontinence episodes and quality of life surveys.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Stress Urinary Incontinence symptoms
* Urodynamic stress incontinence confirmed with multichannel urodynamic testing
* positive cough stress test
* urgency score < stress score
* Patient's age between 40 - 65 years
* Desire to surgical correction of stress urinary incontinence or inadequate response to conservative treatment of SUI

Exclusion Criteria:

* Post-void residual volume >100cc
* Detrusor overactivity on preoperative multichannel urodynamic testing
* History of previous synthetic, biologic or fascial sub-urethral sling or any other surgery on external genitalia, bladder neck, bladder or urethra
* Desires future childbearing
* Chronic inguinal or vulvar abscess or history of Hidradenitis Suppurative
* History of bleeding diathesis or current anti-coagulation therapy
* Inguinal lymphadenopathy or inguinal/vulvar mass
* Current genitourinary fistula or urethral diverticulum
* Current sever cystocele or rectocele
* Active urinary infection
* Non-treated urge incontinency or any significant voiding dysfunction
* Neuromuscular disorders
* Uncontrolled Diabetes
* Reversible cause of incontinence (i.e. drug effect)
* Contraindications for surgery

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
24hours voiding diary reduction | 1month
  Evaluation the 24hours voiding diary reduction by patient questionaire 2h pad test and By clinical measures by cystourethroscopy and urodynamic before , 1, 3,6 and 12 months after MDCs injection.

SECONDARY OUTCOMES:
Enhance incontinence quality of life (I-Qol) | 1 month
  Evaluation the enhance incontinence quality of life (I-Qol) by questionnaire form, before injection of MDCs, 1, 3,6 and 12 months after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Department of Regenerative Medicine And Royan Cell Therapy Center Royan Institute For stem Cell Biology and Technology; Farzaneh Sharifiaghdas, MD, Study Director — Urology and Nephrology Research Center, Shahid Beheshti University; Reza Moghadasali, PhD, Principal Investigator — Department of Regenerative Medicine And Royan Cell Therapy Center Royan Institute For stem Cell Biology and Technology; Farzam Tajali, MD, Principal Investigator — Urology and Nephrology Research Center, Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.org